CLINICAL TRIAL: NCT02235584
Title: Loss of Insulinotropic Properties of Glucagon-like Peptide-1 (GLP-1) and Glucose-dependent Insulinotropic Peptide (GIP) After Glucocorticoid Induced Insulin Resistance
Brief Title: Insulinotropic Effect of GLP-1 and GIP After Dexamethasone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Carsten Dirksen, MD, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-D-2009-070
Record Dates: First submitted 2014-09-07; First posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Type 2 Diabetes
Keywords: Incretin hormones; GLP-1; GIP; Dexamethasone
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexamethasone (Experimental): This is a before-after study. All subjects are administered dexamethasone 2mg BID for 5 days.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone are given dexamethasone tablets of 2mg twice daily.

SUMMARY:
In this study we examine whether inducing insulin resistance by dexamethasone in healthy volunteers will lead to a decreased insulinotropic effect of the hormones GLP-1 and GIP.

DETAILED DESCRIPTION:
In this study we are going to examine the insulinotropic properties of GLP-1 and GIP before and after the development of insulin resistance and/or glucose intolerance.The insulinotropic properties of GLP-1 and GIP are greatly reduced in type 2 diabetes.

Since the development of type 2 diabetes is preceded by insulin resistance and glucose intolerance we wanted to examine the insulinotropic properties of GLP-1 and GIP in the early stages of type 2 diabetes.

To do this, we want to induce insulin resistance and/or glucose intolerance. This is achieved by 5 days of treatment with dexamethasone.

Subjects are studied on 4 different days in randomized order, with an oral glucose tolerance test (OGTT) and glucose clamps + infusions of GLP-1, GIP and NaCl before and immediately after 5 days treatment with dexamethasone, 2mg bid. On day 1, 2 and 3 after the 5 days of dexamethasone, 2mg dexamethasone was given in the afternoon after the tests to ensure unchanged insulin resistance

ELIGIBILITY:
Inclusion Criteria:

* Caucasians above 20 and below 45 years of age
* Normal glucose tolerance as assessed by the WHO criteria
* First degree relative and at least 1 second degree relative with type 2 diabetes
* Normal haemoglobin
* Informed consent

Exclusion Criteria:

* Liver disease (ALAT/ASAT > 2 times normal value)
* Kidney disease (S-creatinin > 130uM and/or albuminuria)
* Heart disease (NYHA II, III or IV)
* Treatment with medicine that cannot be paused
* Pregnancy of breast feeding

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2009-07; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The potentiating effects of GLP-1 on second phase insulin response when clamped at at bloodsugar of 7 mmol/l | 1-3 days after dexamethasone treatment
  After dexamethasone treatment subjects are tested with infusion of GLP-1 during a clamped blood-sugar of 7mmol/l. Their increase in the second phase insulin response is the primary endpoint.

SECONDARY OUTCOMES:
First phase insulin response to GLP-1 infusion at 7mmol/l | 1-3 days after dexamethasone
First phase insulin response to GIP infusion at 7mmol/l | 1-3 days after dexamethasone
Second phase insulin response to GIP infusion at 7mmol/l | 1-3 days after dexamethasone treatment

OTHER OUTCOMES:
Total insulin response to arginine infusion | 1-3 days after dexamethasone

CONTACTS AND LOCATIONS:
Overall Officials: Thure Krarup, dr. med., Study Director — Bispebjerg Hospital
Locations (1):
- Bispebjerg University Hospital, Copenhagen NV, Denmark

REFERENCES:
- [Derived] Eriksen M, Jensen DH, Tribler S, Holst JJ, Madsbad S, Krarup T. Reduction of insulinotropic properties of GLP-1 and GIP after glucocorticoid-induced insulin resistance. Diabetologia. 2015 May;58(5):920-8. doi: 10.1007/s00125-015-3522-y. Epub 2015 Mar 9. PMID 25748606